CLINICAL TRIAL: NCT02971891
Title: A Phase 3, Randomized, Double-Blind, Vehicle-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of CLS006 Versus Vehicle in Subjects 2 Years of Age or Older With Cutaneous Common Warts
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of CLS006 Versus Vehicle in Subjects 2 Years of Age or Older With Cutaneous Common Warts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLS006-CO-PR-001
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Cutaneous Common Warts
MeSH Terms: interventions — Furosemide; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- CLS006 (Furosemide) (Experimental): CLS006 (Furosemide) Topical Gel, 0.125%
  Interventions: Drug: CLS006 (Furosemide) Topical Gel
- Vehicle (Placebo Comparator): Vehicle Topical Gel
  Interventions: Drug: Vehicle Topical Gel

INTERVENTIONS:
Drug: CLS006 (Furosemide) Topical Gel
  Arms: CLS006 (Furosemide)
Drug: Vehicle Topical Gel
  Arms: Vehicle

SUMMARY:
To evaluate the efficacy and safety of six (6) weeks of once daily application of Furosemide Topical Gel 0.125% (CLS006) compared to vehicle in subjects ≥ 2 years of age with nongenital cutaneous common warts (verruca vulgaris).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have 1 to 6 clearly identifiable common warts located on hands feet limbs, and/or trunk

  * Each wart must measure 3 to 10 mm in their longest dimension (diameter) on the epidermal plane of the skin at baseline visit,
  * Each wart must be present for at least 4 weeks at the baseline visit,
  * Plantar, facial, subungual, and common warts in regions of a pre-existing inflammatory condition are excluded. In addition, other warts (e.g., flat, genital) are excluded.
* Male or female subjects 2 years of age or older
* Females of childbearing potential who are using a highly effective form of birth control or females of non-childbearing potential
* Negative in-office urine pregnancy test at Screening and Baseline
* Subjects free of any clinically significant dermatologic disorder in the treatment area
* Subjects free of any clinically significant systemic condition which will interfere with the study assessments or increase the risk of AEs
* Subjects willing to refrain from using other topical products in the treatment area, or prohibited medications for the duration of the study

Exclusion Criteria:

* Subjects who have used any wart treatments/therapies, prescription or over-the-counter, as follows:

  * Salicylic acid, cantharidin, sinecatechins (VeregenTM), simple occlusion (e.g., duct tape), and/or any other over-the-counter wart-removing products in the treatment area within 4 weeks of the Baseline Visit.
  * Cryotherapy (e.g., treatment with liquid nitrogen), carbon dioxide, electrodessication, laser, surgery, or other forms of mechanical destruction (e.g., emery boards, clippers, debriders, etc.) in the treatment area within 8 weeks of the Baseline Visit.
  * Treatment with immunotherapy (DPCP, DNCB or other), imiquimod, 5-fluorouracil,bleomycin, podophyllin or any other wart immunotherapy or treatment (e.g., Candida antigen) designed to stimulate immune response within 12 weeks of the Baseline Visit.
* Subjects who are immunocompromised.
* Subjects who have taken, within 30 days prior to the Baseline visit, or require treatment with systemic immunosuppressive or immunomodulatory medication (including oral or parenteral corticosteroids) during the course of the study
* Subjects who require ongoing treatment with oral or injectable furosemide
* Subjects who have used an investigational drug/device within 30 days of the Baseline visit
* Subjects with known sensitivities to any of the investigational product ingredients including furosemide (or other sulfonamides).
* Subjects who have a clinically significant abnormality of the cardiovascular, hepatic or renal systems.
* Subjects with clinically relevant/significant abnormal laboratory results, vital signs, ECG, and/or physical findings at Screening and/or Baseline
* Subjects with a chronic medical condition or clinically significant abnormal physical or laboratory finding(s) that may require the use of a prohibited medication/treatment.
* Subjects who currently abuse alcohol or drugs or who have a history of chronic alcohol or drug abuse within the past year.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2017-01; Primary Completion 2018-04-16 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Mobile, Alabama
  - Glendale, Arizona
  - Los Angeles, California
  - Santa Monica, California
  - Santa Rosa, California
  - Denver, Colorado
  - Miami, Florida
  - North Miami Beach, Florida
  - Ormond Beach, Florida
  - Tampa, Florida
  - Plainfield, Indiana
  - Lake Charles, Louisiana
  - Monroe, Louisiana
  - Hunt Valley, Maryland
  - Beverly, Massachusetts
  - Fort Gratiot, Michigan
  - Omaha, Nebraska
  - Portsmouth, New Hampshire
  - New York, New York
  - High Point, North Carolina
  - Wilmington, North Carolina
  - Fort Washington, Pennsylvania
  - Hazleton, Pennsylvania
  - Austin, Texas
  - College Station, Texas
  - Katy, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects must have 1 to 6 clearly identifiable common warts located on hands, feet, limbs, and/or trunk
Groups:
- CLS006 (Furosemide): CLS006 (Furosemide) Topical Gel applied once daily CLS006 (Furosemide) Topical Gel, 0.125%
- Vehicle: Vehicle Topical Gel applied once daily Vehicle Topical Gel
Period: Overall Study
Arm/Group | CLS006 (Furosemide) | Vehicle
Started | 246 | 238
Subjects Who Had 1 Wart | 118 | 117
Subjects Who Had 2 Warts | 56 | 53
Subjects Who Had 3 Warts | 24 | 24
Subjects Who Had 4 Warts | 21 | 12
Subjects Who Had 5 Warts | 12 | 11
Subjects Who Had 6 Warts | 15 | 21
Completed | 229 | 214
Not Completed | 17 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CLS006 (Furosemide) | Vehicle | Total
Number analyzed (Participants) | 246 | 238 | 484
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (16.40) | 29.1 (16.57) | 28.8 (16.47)
Age, Customized [Count of Participants; unit: Participants]
  >=2 to <12 | 43 | 37 | 80
  >=12 to <18 | 41 | 43 | 84
  >=18 to <65 | 158 | 154 | 312
  >=65 | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 101 | 206
  Male | 141 | 137 | 278
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 39 | 78
  Not Hispanic or Latino | 205 | 199 | 404
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 12 | 10 | 22
  White | 226 | 221 | 447
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Proportion of Subjects With Complete Clearance of All Treated Warts Between the Active and Vehicle at Week 18/End of Post-treatment Efficacy Evaluation.
Time Frame: Week 18
Measure: Count of Participants; unit: Participants
Arm/Group | CLS006 (Furosemide) | Vehicle
Number analyzed (Participants) | 229 | 214
Participants
  Achieved complete clearance of all treated warts | 32 | 24
  Not achieved complete clearance of all treated warts | 197 | 190
Statistical Analysis 1: Comparison: CLS006 (Furosemide); Test type: Superiority; p = 0.1789, Cochran-Mantel-Haenszel

2. Secondary Outcome: The Ratio of the Number of Cleared Warts Out of the Number of Treated Warts for Each Subject
Time Frame: Week 18
Measure: Mean (Standard Deviation); unit: ratio of cleared warts
Arm/Group | CLS006 (Furosemide) | Vehicle
Number analyzed (Participants) | 229 | 214
ratio of cleared warts | 0.178 (0.3636) | 0.145 (0.3334)

3. Secondary Outcome: Difference in the Proportion of Subjects With Complete Clearance of All Treated Warts at Week 12.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | CLS006 (Furosemide) | Vehicle
Number analyzed (Participants) | 229 | 214
Participants
  Complete clearance of all treated warts | 21 | 14
  Not complete clearance of all treated warts | 208 | 200

4. Secondary Outcome: The Ratio of Cleared Warts to All Treated Warts for Each Subject at Week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: ratio of cleared warts
Arm/Group | CLS006 (Furosemide) | Vehicle
Number analyzed (Participants) | 229 | 214
ratio of cleared warts | 0.120 (0.3041) | 0.087 (0.2601)

5. Secondary Outcome: Change From Baseline in Wart Size for Each Subject
Time Frame: Week 18
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CLS006 (Furosemide) | Vehicle
Number analyzed (Participants) | 229 | 214
mm | -2.5 (7.13) | -2.4 (6.64)

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | CLS006 (Furosemide) | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/246 | 0/238
Serious Adverse Events (participants affected / at risk) | 0/246 | 0/238
Other Adverse Events (participants affected / at risk) | 9/246 | 9/238
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CLS006 (Furosemide) (N=246) | Vehicle (N=238)
Upper respiratory tract infection (Infections and infestations) | 5 | 2
Headache (Nervous system disorders) | 3 | 3
Sinusitis (Infections and infestations) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT02971891/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT02971891/SAP_001.pdf